CLINICAL TRIAL: NCT04785014
Title: Effect of USG-guided Baker's Cyst Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, nurmuhammet tas, phd, Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ErzurumRTRHh
Record Dates: First submitted 2021-02-25; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Baker Cyst; Knee Disease
Keywords: Baker's cyst; Ultrasonography,; Cyst aspiration; Knee exercises for Baker's cyst; Cold pack
MeSH Terms: conditions — Popliteal Cyst | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspiration group (Experimental): In the aspirated group, the popliteal fossa areas were sterilized and BC content was aspirated from the popliteal fossa percutaneously under USG guidance with a 21-gauge needle (Figure 1). If the BC was septal, aspiration was performed from several different levels of the cyst so that the cyst content could be completely emptied.Additionally, the participants in both groups were trained on how to perform exercises and were also recommended to practice cold treatment for 15 min both in the morning and evening for 2 weeks.
  Interventions: Procedure: interventional
- control group (Active Comparator): no aspiration was performed in the control group. Additionally, the participants in both groups were trained on how to perform exercises and were also recommended to practice cold treatment for 15 min both in the morning and evening for 2 weeks.
  Interventions: Procedure: interventional

INTERVENTIONS:
Procedure: interventional — In the aspirated group, the popliteal fossa areas were sterilized and BC content was aspirated from the popliteal fossa percutaneously under USG guidance with a 21-gauge needle (Figure 1). If the BC was septal, aspiration was performed from several different levels of the cyst so that the cyst content could be completely emptied.

SUMMARY:
ABSTRACT Objective: The aim of this study was to investigate the effect of ultrasonography (USG)-guided Baker's cyst (BC) aspiration in the treatment of BC.

Design: A total of 40 patients presented to our polyclinic with the complaints of swelling at the back of the knee. The 40 patients were randomly divided into two groups: (I) aspiration group (n=20) and (II) control group (n=20). In the aspiration group, BC content was aspirated percutaneously under USG guidance, whereas no aspiration was performed in the control group. Additionally, the participants in both groups were trained on how to perform exercises and were also recommended to practice cold treatment for 15 min both in the morning and evening for 2 weeks. All the patients were followed up with USG at the first and third months, VAS, WOMAC, NHP , Lysholm and Cincinnati. The success of the treatment was demonstrated by the decrease in the width, length and area of the BCs and Lysholm, Cincinnati ,VAS, WOMAC and NHP scores.

DETAILED DESCRIPTION:
Objective: The aim of this study was to investigate the effect of ultrasonography (USG)-guided Baker's cyst (BC) aspiration in the treatment of BC.

Design: This prospective study was conducted at Erzurum Atatürk University Medical Faculty Physical Medicine and Rehabilitation Department between January 2016 and June 2017 for a total period of 18 months. A total of 40 patients (11 males, 29 females) aged between 33-71 (mean age, 55.9 ± 9.6) years presented to our polyclinic with the complaints of swelling at the back of the knee. All the patients signed an informed consent form and the study was approved by the local ethics committee. (ERZURUM ATATUK UNIVERSITY MEDICAL FACULTY CLINICAL RESEARCH ETHICS COMMITTEE Date:03.12.2015 Meeting Number:8 Decision Number:24) Patients with a history of malignancy, coagulation disorder, and a neurological deficit and those receiving anticoagulant therapy were excluded from the study. The sample size was determined with a 95% confidence interval according to https://www.macorr.com/sample-size-calculator.htm website.

Prior to the procedure, all the patients were evaluated with grey-scale USG using an Esaote MyLab 60 USG device with a linear probe of 7.5 MHz. On USG examination, the area of transverse diameter(width-parallel to the knee joint), longitudinal diameter (length-perpendicular to the knee joint), and the USG area( from the widest place viewed) of BCs were calculated and recorded.

Clinical complaints of the patients, long-term complaints, and the history of medical, interventional, and surgical treatments were reviewed for each patient. Patients were also investigated for acute local or systemic infections.

The severity of clinical complaints was assessed using VAS, WOMAC knee osteoarthritis index, Lysholm knee scoring scale, Cincinnati knee rating system, and NHP. Patients with BC who had no contraindications for treatment and completed the WOMAC Knee osteoarthritis index, Lysholm knee scoring scale, Cincinnati knee rating system, VAS, and NHP and signed the patient consent form were included in the study. Patients were randomly divided into two groups by consecutive alternate allocation according to the time of admittance: (I) aspiration group (n=20) included the patients aspirated and (II) control group (n=20) included those who did not aspirated. In the aspirated group, the popliteal fossa areas were sterilized and BC content was aspirated from the popliteal fossa percutaneously under USG guidance with a 21-gauge needle (Figure 1). If the BC was septal, aspiration was performed from several different levels of the cyst so that the cyst content could be completely emptied. In contrast, no aspiration was performed in the control group. Additionally, the participants in both groups were trained on how to perform exercises and were also recommended to practice cold treatment for 15 min both in the morning and evening for 2 weeks.

After the aspiration, the patients were told how to exercise and practice cold treatment in the morning and evening for 2 weeks. Patients were discharged after a 30-min observation period following the procedure. Patients were allowed to apply bandages for 2 days after the procedure and were followed pre- and post-procedurally at the first and third months of treatment with WOMAC Knee osteoarthritis index, Lysholm knee scoring scale, Cincinnati knee rating system, VAS, and NHP and with USG. The appearance of BC at month 3 was examined on grey-scale USG and the length, width, and area of the cyst were recalculated. During the 3-month follow-up period, no additional treatment was performed in any patient. The success of the procedure was defined as reduction in BC width, length and area in sonographic measurements and decrease in the Lysholm knee scoring scale, Cincinnati knee rating system, VAS, WOMAC knee osteoarthritis index, and NHP scores.

ELIGIBILITY:
Inclusion Criteria:

* To have baker's cyst..
* To comply with the treatment protocol
* Signing the information consent form

Exclusion Criteria:

* To have malignancy
* To have neurological deficit
* Those with coagulation disorders or those receiving anticoagulant therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Effect of USG-guided Baker's cyst aspiration | 12 week
  Baker's cyst USG measurement width:mm
Effect of USG-guided Baker's cyst aspiration | 12 week
  Baker's cyst USG measurement length:mm
Effect of USG-guided Baker's cyst aspiration | 12 week
  Baker's cyst USG measurement area:mm^2
Effect of USG-guided Baker's cyst aspiration | 12week
  Visual Analog Score for pain
Effect of USG-guided Baker's cyst aspiration | 12week
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) for Pain,Stiffness, and Physical Function .The minimum and maximum values respectively 0/96 and higher scores mean a worse outcome
Effect of USG-guided Baker's cyst aspiration | 12week
  Nottingham Health Profile (NHP) for quality of life .The minimum and maximum values respectively 0/600 and higher scores mean a worse outcome
Effect of USG-guided Baker's cyst aspiration | 12week
  Tegner Lysholm Knee Scoring Scale for how your knee pain has affected your ability to manage in everyday life. .The minimum and maximum values respectively 0/100 and higher scores mean a better outcome
Effect of USG-guided Baker's cyst aspiration | 12week
  Cincinnati Knee Rating System score for a variety of symptoms, sports and daily activity functions, and objective physical findings.The minimum and maximum values respectively 0/30 and higher scores mean a better outcome

IPD SHARING:
Plan to Share IPD: Yes
: A total of 40 patients presented to our polyclinic with the complaints of swelling at the back of the knee. The 40 patients were randomly divided into two groups: (I) aspiration group (n=20) and (II) control group (n=20). In the aspiration group, BC content was aspirated percutaneously under USG guidance, whereas no aspiration was performed in the control group. Additionally, the participants in both groups were trained on how to perform exercises and were also recommended to practice cold treatment for 15 min both in the morning and evening for 2 weeks. All the patients were followed up with USG at the first and third months, VAS, WOMAC, NHP , Lysholm and Cincinnati. The success of the treatment was demonstrated by the decrease in the width, length and area of the BCs and Lysholm, Cincinnati ,VAS, WOMAC and NHP scores.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This prospective study was conducted at Erzurum Atatürk University Medical Faculty Physical Medicine and Rehabilitation Department between January 2016 and June 2017 for a total period of 18 months.
Access Criteria: To all researchers..